CLINICAL TRIAL: NCT07297134
Title: Serum PTEN Levels and Organ-Specific microRNA Signatures as Predictors of Metastatic Patterns in Breast Cancer: A Prospective Observational Study
Brief Title: PTEN and Organ-Specific microRNAs in Metastatic Breast Cancer
Acronym: PTEN-miR-MBC
Status: Recruiting | Type: Observational
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Emine YILDIRIM, associate professor, MD, Atlas University
Other Study IDs: MBC-PTEN-miRNA
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Metastatic Breast Cancer; miRNAs; PTEN
Keywords: Breast Cancer; Metastatic Breast Cancer; miRNAs; PTEN; Breast Cancer Biomarkers; Organ Specific Metastasis; miRNA Profiling
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples collected during routine venous blood draws for PTEN quantification and microRNA profiling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Metastatic Breast Cancer: Participants diagnosed with breast cancer and radiologically confirmed distant metastasis to bone, liver, lung, or brain.
- Non-Metastatic Early-Stage Breast Cancer: Participants diagnosed with early-stage and local advenced (Stage I-III) breast cancer with no clinical or radiological evidence of distant metastasis.
- Healthy Controls: Age-matched healthy individuals without known malignancy or active systemic disease.

SUMMARY:
This prospective observational study aims to evaluate serum levels of PTEN, a tumor suppressor gene, and organ-specific microRNAs (miRNAs) associated with metastatic patterns in breast cancer. Serum samples will be analyzed using quantitative reverse transcription polymerase chain reaction (qRT-PCR)-based miRNA profiling and enzyme-linked immunosorbent assay (ELISA)-based PTEN quantification. Three groups will be included: patients with metastatic breast cancer (n=80), patients with non-metastatic early-stage breast cancer (n=40), and healthy controls (n=40).

The primary objective is to identify serum biomarkers that differentiate metastatic from non-metastatic disease. Secondary analyses will evaluate correlations between biomarker levels and organ-specific metastatic involvement, including bone, lung, liver, and brain metastases. Findings from this study may support the development of a noninvasive serum-based tool for predicting metastatic patterns in breast cancer.

DETAILED DESCRIPTION:
Breast cancer is a heterogeneous disease with varying biological behaviors and a strong tendency to metastasize to specific organs, including the bone, liver, lung, and brain. The development of distant metastases remains the primary cause of breast cancer-related mortality. Therefore, the identification of reliable, minimally invasive biomarkers that can predict metastatic spread is a critical unmet clinical need.

MicroRNAs (miRNAs) are small, noncoding RNA molecules that regulate gene expression and have emerged as promising biomarkers due to their stability in the circulation and their association with cancer progression. Specific miRNA expression patterns have been linked to organotropism in breast cancer, including signatures associated with bone, lung, liver, and brain metastases. Additionally, PTEN is a key tumor suppressor gene involved in cell cycle regulation, apoptosis, and PI3K/AKT pathway signaling. Loss of PTEN function is frequently observed in aggressive and metastatic breast cancers, and reduced circulating PTEN levels may correlate with tumor burden and metastatic dissemination.

This prospective observational clinical study aims to evaluate serum PTEN levels and organ-specific miRNA profiles in three participant groups:

Metastatic breast cancer patients (n=80) diagnosed with distant organ involvement.

Early-stage non-metastatic breast cancer patients (n=40) with no radiological or clinical evidence of metastasis.

Healthy control participants (n=40) without known malignancy.

Serum samples will undergo laboratory analysis using two validated molecular techniques:

Quantitative reverse transcription polymerase chain reaction (qRT-PCR) for profiling selected miRNAs associated with organ-specific metastatic patterns.

Enzyme-linked immunosorbent assay (ELISA) for quantification of circulating PTEN protein levels.

The primary objective of the study is to compare serum PTEN and miRNA expression levels between metastatic and non-metastatic breast cancer groups, as well as healthy controls. Secondary objectives include assessing associations between these biomarkers and (a) the number of metastatic sites, (b) specific organ involvement (bone, lung, liver, brain), and (c) selected clinical characteristics, including hormone receptor status, HER2 expression, patient age, and stage at diagnosis.

The overarching goal is to characterize a panel of circulating biomarkers that may contribute to early detection of metastatic potential and organ-specific metastatic patterns in breast cancer. Identifying such signatures may facilitate noninvasive risk stratification, support personalized treatment planning, and form the basis for future translational research aimed at developing clinically applicable diagnostic assay

ELIGIBILITY:
Inclusion Criteria:

* Female individuals aged ≥18 years
* Ability to provide written informed consent
* Group I (Metastatic BC): Histopathologically confirmed breast cancer and radiologically or clinically proven distant organ metastasis at the time of enrollment
* Group II (Non-Metastatic BC): Histopathologically confirmed breast cancer with no evidence of distant metastasis
* Group III (Healthy Controls): Women ≥18 years with no known breast disease and no personal history of malignancy

Exclusion Criteria:

* History of any other primary malignancy
* Known breast disease or breast cancer diagnosis in Group III
* Immunosuppressive therapy that may alter immune or biomarker profiles
* Active infection or inflammatory condition that may alter biomarker levels
* Inability or unwillingness to provide informed consent
* Severe hepatic, renal, or hematologic dysfunction
* Current pregnancy or lactation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three groups were included in this study: women with metastatic breast cancer, women with early or locally advanced nonmetastatic breast cancer, and age-matched healthy female controls.
  Participants in the metastatic group have radiologically or clinically confirmed distant organ involvement. The nonmetastatic group includes patients with histopathologically confirmed breast cancer without any evidence of distant metastasis. Healthy controls consist of women without known breast disease, malignancy, or systemic illness. All participants are aged 18 years or older and able to provide informed consent. Recruitment will occur through oncology clinics, breast surgery units, and outpatient services.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Serum PTEN Level | At enrollment (single blood draw)
  Quantification of circulating PTEN protein levels in serum using enzyme-linked immunosorbent assay (ELISA) and comparison between metastatic breast cancer, non-metastatic breast cancer, and healthy control groups.
Serum microRNA (miRNA) Expression Levels | At enrollment
  Expression levels of selected organ-specific microRNAs (bone, lung, liver, and brain associated miRNAs) measured by qRT-PCR in all study groups.

SECONDARY OUTCOMES:
Correlation Between Biomarker Levels and Metastatic Organ Involvement | At enrollment
  Correlation of serum PTEN and miRNA expression levels with the presence of metastasis in specific organs (bone, liver, lung, brain).
Comparison of Biomarker Levels Between Single-Organ and Multi-Organ Metastasis | At enrollment
  Comparison of serum PTEN and miRNA levels between patients with single-site metastasis and those with multi-site metastases.
Correlation Between Biomarkers and Clinical Variables | At enrollment
  Exploratory analysis evaluating correlation between serum PTEN/miRNA levels and clinical features including hormone receptor status (ER/PR), HER2 status, age, tumor stage, and grade

CONTACTS AND LOCATIONS:
Locations (1):
- Atlas University Faculty of Medicine, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy and data protection regulations. Only de-identified, aggregate results may be shared with researchers upon reasonable request.